CLINICAL TRIAL: NCT05467618
Title: Comparison of Intra-oral and Extra-oral Surgical Approach in Reducing Fractures at the Angle of the Mandible
Brief Title: Comparison of Surgical Approaches in Reducing Mandibular Angle Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayub Teaching Hospital (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Principal Investigator, Shahid ali shah, Assistant Professor, Ayub Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sashah0001
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Fractures, Bone; Mandibular Fractures
MeSH Terms: conditions — Fractures, Bone; Mandibular Fractures | interventions — Surgery, Oral

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with non-probability consecutive sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-Oral Surgical approach (Experimental): The mandibular fracture was reduced using an intra-oral surgical approach.
  Interventions: Procedure: Maxillofacial surgery
- Extra-Oral Surgical approach (Experimental): An External/Facial approach was used to reduce the mandibular bone fracture.
  Interventions: Procedure: Maxillofacial surgery

INTERVENTIONS:
Procedure: Maxillofacial surgery — An incision on the skin over the mandible versus incision on the gingivae inside the mouth

SUMMARY:
This study compared the surgical approach to the lower jaw fractures, an approach from the face and an approach from inside the mouth were used and compared for the outcomes.

DETAILED DESCRIPTION:
Mandibular factures tend to be more common than those of the middle third of the face.1 They occur alone or in combination with other facial bone fractures resulting in severe loss of function and disfigurement.2,3 Mandibular factures tend to be more common than those of the middle third of the face.1 They occur alone or in combination with other facial bone fractures resulting in severe loss of function and disfigurement.2,3 The pattern of mandibular fractures varies with geographic location, physical activity, social, cultural and environmental factors. The main causes 4,5 of mandibular fracture are; Road traffic accidents, interpersonal violence, falls, sports injuries, industrial trauma, pathological fractures etc. In developing countries road traffic accident 6 is the common cause of mandibular fractures due to lack of implementation of traffic laws while in developing countries alcohol related7 interpersonal violence is the leading cause. Any age and sex group may sustain trauma to the lower jaw but children below the age of 12 years are less susceptible to fracture because their bones are more resilient.5,6 Different modalities available for the treatment of mandibular fractures are: Maxillo mandibular fixation (MMF) alone e.g. dental wiring, arch bar etc.8 Previously traditional methods i.e. maxillomandibular fixation and transosseous wiring were the most popular methods used for mandibular fracture fixation. These are still commonly used methods9 and have got various disadvantages such as preventing normal jaw function, weight loss due to restriction of food to liquid consistency, oral hygiene problem and reduction of ventilatory volume.,10 Currently, fixation with one or two mini- plates has become a widely acceptable method of providing internal fixation and eliminating the need for post-operative maxillo mandibular fixation. The fixation of mandibular angle can be carried out by two methods i.e. Intra oral approach8, and Extra oral approach. For intra oral approach buccal sulcus incision while for extra oral approach sub-mandibular (Risdon),11 incision is given. Postoperative complications related to both types of treatment modalities were observed in intra oral approach 13.3 % and extra oral approach 16.6% infection and limited opening were observed in intra oral approach 6.6% and extra oral approach 16.6%.12 Rationale of this study is to compare post-operative complication of intra oral approach and extra oral approach in reduction of mandibular angle fracture in terms of infection and limited mouth opening. In our study, if we find less complication of intra-oral approach in significant number of patients, we will strongly recommend its routine use in the reduction of pain and limited mouth opening.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 16 to 60 years
* Both Genders.
* Patients undergoing surgery for mandibular angle fracture

Exclusion Criteria:

* Pathological fractures.
* Condylar and sub-condylar fractures.
* Edentulous patients.
* Fire arm injury (FAI).
* Fractures of the middle third of face.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Indication of post-surgical infections | Up to three weeks
  Redness, swelling, pain, bleeding, or any discharge
Limited jaw opening | Up to three weeks
  Mouth opening considered limited if the patient can only open mouth to a width of less than the width of his/her three fingers (index, middle, ring).

CONTACTS AND LOCATIONS:
Overall Officials: Alman Khan, BDS,FCPS, Principal Investigator — Ayub Teaching Hospital
Locations (1):
- Ayub Teaching Hospital, Abbottābād, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
These are walk-in patients to the facility and we are officially obligated to keep their confidentiality. The facility may be approached for the data and data maybe provided subject to the approval of the subjects.

REFERENCES:
- [Background] 1. Abbas I, Ali K. Management of mandibular fractures a prospective study; Pak Oral Dent 2007;22:151-2.
- [Background] 2. Muzzafar K. Management of maxillofacial trauma. AFID Dent J 2008;10:18-21.
- [Background] 3. Nayyak MS, Ekanayake MBK. Assessment of maxillofacial injuries. Pakistan Oral Dent J 2007;21:12-8.
- [Background] Abbas I, Ali K, Mirza YB. Spectrum of mandibular fractures at a tertiary care dental hospital in Lahore. J Ayub Med Coll Abbottabad. 2003 Apr-Jun;15(2):12-4. PMID 14552240
- [Background] 5. Zaki MA, Islam T, Mamon S, Aleem A. Pattern of maxillofacial injuries received at Abassi Shaheed Hospital, KMDC, Karachi. Annual Abassi Shaheed Hosp. 2008;7:291-3.
- [Background] Lawoyin DO, Lawoyin JO, Lawoyin TO. Fractures of the facial skeleton in Tabuk North West Armed Forces Hospital: a five year review. Afr J Med Med Sci. 1996 Dec;25(4):385-7. PMID 9532313
- [Background] Edwards TJ, David DJ, Simpson DA, Abbott AA. Patterns of mandibular fractures in Adelaide, South Australia. Aust N Z J Surg. 1994 May;64(5):307-11. doi: 10.1111/j.1445-2197.1994.tb02216.x. PMID 8179524
- [Background] 8. Patel MF. Fixation techniques & mandibular osteosynthesis. In: Langdon JD, Patel MF. Operative maxillofacial surgery. 1st ed London: Chapman & Hall, 2005;331-45.
- [Background] Renton TF, Wiesenfeld D. Mandibular fracture osteosynthesis: a comparison of three techniques. Br J Oral Maxillofac Surg. 1996 Apr;34(2):166-73. doi: 10.1016/s0266-4356(96)90372-1. PMID 8861293
- [Background] Moreno JC, Fernandez A, Ortiz JA, Montalvo JJ. Complication rates associated with different treatments for mandibular fractures. J Oral Maxillofac Surg. 2000 Mar;58(3):273-80; discussion 280-1. doi: 10.1016/s0278-2391(00)90051-x. PMID 10716108
- [Background] 11. Risdon F: Ankylosis of Temporomandibular Joint. J Am Dent Assoc 2008; 21:1933.
- [Background] 12. Ali S, Warraich A. Comparison of two surgical procedures in reduction of mandibular angle fracture. Pak oral Dent J. 2010;30(2):287-90.